CLINICAL TRIAL: NCT01442753
Title: Family-Skills Training to Prevent Tobacco and Other Substance Use in Latino Youth: A CBPR RCT
Brief Title: Family-Skills Training to Prevent Tobacco and Other Substance Use in Latino Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2010NTLS088; 1008S86938 (Other: IRB, University of Minnesota); 1U54CA153603-01 (NIH)
Record Dates: First submitted 2011-09-19; First posted 2011-09-29 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Tobacco Use Disorder; Alcohol Use Disorder; Drug Use Disorder; Smoking; Alcohol Drinking; Drug Abuse
Keywords: Spanish speaking
MeSH Terms: conditions — Tobacco Use Disorder; Alcoholism; Substance-Related Disorders; Smoking; Alcohol Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Active Comparator): Families will be randomized to either receive the intervention (family-skills training) immediately. The intervention will be delivered over eight weeks. Sessions will be divided between self-reflection, didactics, and skill-building exercises all aimed at developing strong parenting practices and facilitating relationship building between parents and youth.
  Interventions: Behavioral: Family-Skills Training
- Control Group (Active Comparator): Control group will receive the intervention (family-skills training) in approximately ten months. The intervention will be delivered over eight weeks. Sessions will be divided between self-reflection, didactics, and skill-building exercises all aimed at developing strong parenting practices and facilitating relationship building between parents and youth.
  Interventions: Behavioral: Family-Skills Training

INTERVENTIONS:
Behavioral: Family-Skills Training — Sessions will be divided between self-reflection, didactics, and skill-building exercises all aimed at developing strong parenting practices and facilitating relationship building between parents and youth.

SUMMARY:
The goal of this project is to evaluate the effectiveness of a family-based tobacco use prevention intervention directed at immigrant Latino parents of middle school aged youth as delivered in partnership with seven community organizations. The primary outcomes of the study are youth susceptibility to tobacco use, and changes in parenting practices among the parents of the youth. The planning, initiation, and delivery of the intervention will occur in collaboration with community organizations that have identified this project as important to the families they serve. Though the collaboratively designed training curriculum has been successfully tested and a study design for the current project established, a substantive development period for this project will allow the research team and collaborating organizations to consider key aspects of design and delivery.

DETAILED DESCRIPTION:
This study design is a randomized (at the level of the family) controlled trial (RCT), with a delayed treatment condition for the control group. Participants will be enrolled from community agencies known and trusted within the Latino community including two clinics, a school, three social service agencies and a University of Minnesota Extension site that are likely end-users of the intervention programming.

ELIGIBILITY:
Inclusion Criteria:

* Parent Inclusion

  * Either mother or father born in Latin American country
  * Speaks Spanish
  * Parent willing to give consent for self & youth
* Youth Inclusion

  * Age 10-14 years
  * Speak English or Spanish
  * Youth willing to give assent

Exclusion Criteria:

* Parent Exclusion

  * Not meeting inclusion criteria
  * Past participant Padres Informados parenting program

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2011-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Comparison of susceptibility rate differences between the control and intervention groups | 6 Months Post Intervention
  Youth tobacco use intentions, Questions are 1) "Do you think you will try a cigarette soon?' (not asked of puffers), 2) "Do you think you will be smoking cigarettes one year from now?", and 3) "If one of your best friends were to offer you a cigarette, would you smoke it?" A never-smoker will be considered non-susceptible if answer to the first question is 'No' and answers to both questions 2 and 3 are 'Definitely not'; a puffer will be considered non-susceptible if answers to questions 2 and 3 are 'Definitely not'.

SECONDARY OUTCOMES:
Effect of a family-based intervention | 6 Months
  Parenting behaviors - Monitoring knowledge: child disclosure, parental solicitation and control. Personal involvement: measures parent behavior indicative of their efforts to be aware of adolescents' activities and experiences. Consistent discipline: scale based on work conducted at the ASU Prevention Research Center. Self-efficacy - parent perceives him/herself capable of performing behaviors instrumental to good parenting practice/good developmental outcomes for their children. Social Support: The MSPSS101 measures perceived support from 3 domains: family, friends, and significant other.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Allen, M.D., Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Allen ML, Hurtado GA, Garcia-Huidobro D, Davey C, Forster J, Reynoso U, Alvarez de Davila S, Linares R, Gonzales N, Veronica Svetaz M. Cultural Contributors to Smoking Susceptibility Outcomes Among Latino Youth: The Padres Informados/Jovenes Preparados Participatory Trial. Fam Community Health. 2017 Apr/Jun;40(2):170-179. doi: 10.1097/FCH.0000000000000147. PMID 28207680
- [Derived] Allen ML, Garcia-Huidobro D, Hurtado GA, Allen R, Davey CS, Forster JL, Hurtado M, Lopez-Petrovich K, Marczak M, Reynoso U, Trebs L, Svetaz MV. Immigrant family skills-building to prevent tobacco use in Latino youth: study protocol for a community-based participatory randomized controlled trial. Trials. 2012 Dec 19;13:242. doi: 10.1186/1745-6215-13-242. PMID 23253201